CLINICAL TRIAL: NCT00895219
Title: A Comparison of the Effects of Respiratory Physiotherapy Alone and Respiratory Physiotherapy Combined With Musculoskeletal Techniques in the Management of Dysfunctional Breathing
Brief Title: Physiotherapy and Dysfunctional Breathing
Acronym: HVS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Dr Jennifer A Pryor, Royal Brompton & Harefield NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06/Q0404/64
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-05-08 (Estimated); Status verified 2009-04

CONDITIONS: Hyperventilation
Keywords: Hyperventilation; Dysfunctional breathing; Physiotherapy; Musculoskeletal techniques
MeSH Terms: conditions — Hyperventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Breathing re-training
  Interventions: Other: Breathing re-training
- 2 (Active Comparator): Breathing re-training and musculoskeletal physiotherapy techniques
  Interventions: Other: Breathing re-training and musculoskeletal techniques

INTERVENTIONS:
Other: Breathing re-training — Breathing re-training
  Arms: 1
Other: Breathing re-training and musculoskeletal techniques — Breathing re-training and musculoskeletal physiotherapy techniques including mobilisation techniques to normalise muscle and joint restrictions, doming of the diaphragm to enhance contraction and relaxation, and rib raising to free restriction in rib cage motion.
  Arms: 2

SUMMARY:
Traditionally, the physiotherapy management of people with dysfunctional breathing or hyperventilation syndrome is breathing re-training. There is increasing clinical evidence that structural and functional changes develop in the muscles and connective tissues of the chest wall, abdomen and back when the upper chest accessory pattern of breathing is used over time. When treatment includes breathing techniques only it is difficult for a person with chronic hyperventilation, who has developed muscle and connective tissue changes, to revert to using the normal lower chest diaphragmatic breathing pattern. In clinical practice when the problems which have developed in the musculoskeletal system are addressed, the patient reverts more quickly to the lower chest pattern of breathing but there is as yet little evidence to support this clinical finding.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dysfunctional breathing (Nijmegen score of more than 23)

Exclusion Criteria:

* active metastatic disease
* osteoporotic disease
* dysfunctional breathing as a consequence of respiratory or cardiac disease

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Nijmegen Questionnaire | 0, 2, 4, 8, 12 and 26 weeks

SECONDARY OUTCOMES:
Six-minute walking test | 0, 2, 4, 8, 12 & 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Hodson, MD, Study Director — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton Hospital, London, United Kingdom